CLINICAL TRIAL: NCT00443716
Title: Determination of Adipocyte Parameters in Iliac Crest Biopsies From Post Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-004111; 21b85
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Osteoporosis; Postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: estrogen

SUMMARY:
To evaluate the effect of estrogen treatment on adipocytic and osteoblastic parameters by histomorphometrically measuring adipocyte volume (AV/TV) and adipocyte numbers in goldner's stained iliac crest bone biopsy specimens collected from subjects recruited in the study (IRB number 21B85). The adipocytic parameters will be then correlated with osteoblastic parameters obtained previously during the course of the initai study involving the effect of transdermal estrogen on bone turnover in postmenopausal osteoporotic women.

ELIGIBILITY:
Post-menopausal osteoporotic women

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1985-04; Primary Completion 1989-04 (Actual); Study Completion 1989-04 (Actual)

PRIMARY OUTCOMES:
efficacy of estraderm treatment on osteoporotic women

CONTACTS AND LOCATIONS:
Overall Officials: B. Lawrence Riggs, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States